CLINICAL TRIAL: NCT07155044
Title: Evaluating the Application Value of Neoadjuvant Chemotherapy Compared to Upfront Surgery in Patients With Upper Tract Urothelial Carcinoma
Brief Title: A Comparative Study of Neoadjuvant Chemotherapy Versus Upfront Radical Surgery for Upper Tract Urothelial Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CH-NAC+UTUC
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: UTUC; UC (Urothelial Cancer)
Keywords: NAC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Postoperative pathological tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAC+RNU: Intervention: Participants in this cohort will receive 3-4 cycles of neoadjuvant chemotherapy (NAC) with the gemcitabine and cisplatin (GC) regimen prior to undergoing definitive surgery. Gemcitabine (1000 mg/m²) will be administered on Day 1 and Day 8, and cisplatin (70 mg/m²) will be administered on Day 2 of each 21-day cycle.
  Surgical Intervention: Following the completion of NAC, patients will undergo a radical nephroureterectomy (RNU) with bladder cuff excision. The procedure will be performed via robot-assisted (Da Vinci), laparoscopic, or open approach, based on surgical discretion. Surgery must be performed within 6 weeks (±2 weeks) after the last dose of chemotherapy.
  Objective: The primary objective for this cohort is to evaluate the efficacy of NAC in inducing pathological downstaging (defined as achieving pathological stage <ypT2N0 at surgery) and to assess the pathological complete response (pCR) rate (ypT0N0).
  Interventions: Drug: NAC
- RNU: Intervention: Participants in this cohort will proceed directly to radical nephroureterectomy (RNU) with bladder cuff excision without receiving any prior systemic chemotherapy. The surgery will be scheduled as soon as feasibly possible after enrollment and confirmation of eligibility.
  Surgical Intervention: The surgical approach (robot-assisted, laparoscopic, or open) will be identical to that offered in Cohort A, chosen at the surgeon's discretion based on standard clinical practice.
  Objective: This cohort serves as the control group to provide a contemporary benchmark for standard-of-care outcomes. The objective is to establish the baseline rates of pathological stage distribution, survival, and recurrence without the influence of NAC.

INTERVENTIONS:
Drug: NAC — Participants in NAC+RNU cohort will receive 3-4 cycles of neoadjuvant chemotherapy (NAC) with the gemcitabine and cisplatin (GC) regimen prior to undergoing definitive surgery. Gemcitabine (1000 mg/m²) will be administered on Day 1 and Day 8, and cisplatin (70 mg/m²) will be administered on Day 2 of each 21-day cycle.
  Groups: NAC+RNU

SUMMARY:
This is a single-center, open-label, non-randomized controlled trial comparing the efficacy and safety of neoadjuvant chemotherapy (NAC) followed by radical surgery versus upfront radical surgery alone in patients with high-risk, non-metastatic upper tract urothelial carcinoma (UTUC).

The study aims to answer the following key questions:

Does NAC improve pathologic response rates (defined as downstaging to <ypT2N0) compared to immediate surgery? What is the rate of pathologic complete response (pCR; ypT0N0) in the NAC group? How do the two treatment strategies compare in terms of overall survival, cancer-specific survival, and recurrence-free survival? What is the safety and tolerability profile of NAC using gemcitabine and cisplatin in this patient population? Eligible participants will be assigned to either the NAC-plus-surgery group or the surgery-only group based on clinical evaluation and patient preference. The study will also explore potential biomarkers (e.g., chromosomal instability in liquid biopsies) for predicting treatment response.

Key Eligibility Criteria:

Adults with histologically confirmed high-risk UTUC Clinical stage ≤N1 M0 Adequate renal function (GFR ≥45 mL/min) and ECOG performance status 0-1

Primary Outcome:

Pathologic response rate (proportion of patients with <ypT2N0)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed upper tract urothelial carcinoma (UTUC). For mixed histology, urothelial carcinoma must be the predominant component (≥50%).
* Clinically non-metastatic disease (cN≤1, M0) as determined by cross-sectional imaging (CT or MRI of chest/abdomen/pelvis).
* Planned treatment with radical nephroureterectomy (RNU).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate renal function, defined as glomerular filtration rate (GFR) ≥ 45 mL/min, making the patient a potential candidate for cisplatin-based neoadjuvant chemotherapy.
* Adequate organ and bone marrow function as determined by standard screening tests.
* Recovery from all reversible toxicities of any prior surgery.
* Age ≥ 18 years at the time of enrollment.
* Ability to understand the study and provide signed informed consent.

Exclusion Criteria:

* Radiographic evidence of ≥cN2 lymph node disease or distant metastases (M1).
* History of invasive, lymph node-positive, or metastatic urothelial carcinoma within 2 years prior to enrollment, or history of invasive contralateral UTUC.
* Presence of only a solitary kidney or cisplatin ineligibility.
* Concurrent participation in another interventional clinical trial at the time of enrollment.
* History of a non-urothelial malignant tumor unless the patient has been disease-free for at least 1 year (exceptions include adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix).
* Pregnancy or lactation. Women and men of reproductive potential must agree to use effective contraception.
* Any other medical condition, comorbidity, or psychiatric illness that, in the investigator's judgment, would make the patient an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) with histologically confirmed, non-metastatic upper tract urothelial carcinoma (UTUC) who are planned for radical nephroureterectomy (RNU).
  Participants will be recruited from the urology oncology clinics at a single tertiary care center (e.g., The First Affiliated Hospital of Naval Military Medical University). Eligibility will be determined based on predefined inclusion and exclusion criteria, focusing on patients with adequate renal function (GFR ≥45 mL/min) and performance status (ECOG 0-1) to be potential candidates for cisplatin-based chemotherapy.
  The population will include both patients who are deemed eligible and choose to receive neoadjuvant chemotherapy prior to surgery and those who proceed directly to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Pathological Downstaging Rate (≤ ypT1N0) | Assessed at the time of surgery, approximately 10-14 weeks after initiation of treatment for the NAC+Surgery cohort and approximately 2-4 weeks after enrollment for the Surgery Only cohort.
  The proportion of patients achieving pathological downstaging to stage ≤ ypT1N0 in the surgical specimen following neoadjuvant chemotherapy and radical nephroureterectomy (RNU), as assessed by central pathology review. Patients in the NAC cohort who do not undergo surgery will be classified as non-responders.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Assessed at the time of surgery, approximately 10-14 weeks after initiation of treatment.
  The proportion of patients achieving a pathological complete response (ypT0N0) in the surgical specimen in the NAC+Surgery cohort.
Incidence of Treatment-Related Adverse Events | From start of NAC through surgery (approximately 10-14 weeks).
  Safety and tolerability of neoadjuvant chemotherapy as measured by the incidence, type, and severity of treatment-related adverse events graded according to CTCAE v5.0.
Overall Survival (OS) | From enrollment until death from any cause, assessed up to 60 months.
  The time from the date of enrollment to the date of death due to any cause.
Recurrence-Free Survival (RFS) | From surgery until first documented recurrence or death, assessed up to 60 months.
  The time from surgery to the first documented occurrence of local/regional recurrence, distant metastasis, or death from any cause, whichever occurs first.
Cancer-Specific Survival (CSS) | From enrollment until death due to cancer, assessed up to 60 months.
  The time from enrollment to death directly attributable to upper tract urothelial carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to ensure the confidentiality and privacy of our study participants. The informed consent documents approved by our institutional ethics committee do not include provisions for public sharing of individual-level data. Furthermore, the data contains potentially identifiable sensitive health information, and sharing it would be inconsistent with our commitments to participants and the requirements of local data protection regulations.